CLINICAL TRIAL: NCT00222755
Title: Improving Care for Veterans With Bipolar Disorder
Brief Title: Improving Care for Patients With Bipolar Disorder
Acronym: CIVIC-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Amy Kilbourne, PhD, VA Ann Arbor HCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02394
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2008-01

CONDITIONS: Bipolar Disorder
Keywords: Mood disorders-bipolar; Disease management; Quality of care
MeSH Terms: conditions — Bipolar Disorder | interventions — Disease Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Behavioral Care Management
  Interventions: Behavioral: Disease Management
- 2 (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Disease Management — Self-management, care management, guidelines
  Other Names: Bipolar Care Model
  Arms: 1

SUMMARY:
The purpose of this research study is to learn whether or not a coordinated medical and psychiatric care program can improve outcomes of care for patients with bipolar disorder. We hypothesize that coordinated care via a Care Manager will improve physical and mental health-related quality of life, improve functioning, and reduce symptoms.

DETAILED DESCRIPTION:
Bipolar disorder is a chronic illness associated with significant personal and societal costs. Patients with bipolar disorder also experience more general medical comorbidities than the general population. Potential disparities exist in the receipt of medical and preventive care for individuals with serious mental illness compared to those without serious mental illness. The goal of this study is to pilot test an adapted version of the Wagner Chronic Care Model (CCM). Our target population will be all adult patients with a diagnosis of bipolar disorder (bipolar I, II, NOS) receiving care in the VA Pittsburgh Healthcare System. We plan on consenting and enrolling 60 patients, in which 30 will be randomized to receive the intervention, and 30 will receive usual care. Key components of the intervention include: 1) access to a Care Manager who will help patients make and keep appointments for general medical care by contacting patients on a regular basis; 2) a self-management program, which is education on adherence and self-management for patients by the Care Manager, including information on side-effects, bipolar disorder illness, and tips on communicating with general medical providers that will be provided during group sessions during the first 3 months of the study, and; 3) a registry that tracks patient progress maintained by the Care Manager. Both groups will receive practice guidelines for the treatment of medical conditions tailored to the needs of patients with bipolar disorder. Patients in the intervention arm will meet with the Care Manager after the baseline assessment, who will initially set up regular visits or contacts with the patients and work with them to connect with a primary care clinician. A Survey Coordinator will have patients complete a baseline assessment, and then a follow up assessment at 3 and 6 months later. Our primary outcome is changes in physical and mental health related quality of life. Secondary outcomes include changes in symptoms and functioning. Findings from this study will inform our long-term goal of implementing a larger scale version of the adapted CCM for veterans with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

1. >=18 years old
2. active diagnosis of bipolar disorder
3. have an assigned primary care provider in the VA, and
4. have been seen by a provider in the Beta Team Mood Disorders clinic.

Exclusion Criteria:

1. actively using substances (alcohol or drugs) at the time of enrollment
2. already enrolled in a mental health program with a mobile outreach component in which clinical caregivers deliver services to the patient in the community (e.g., Assertive Community Treatment or Intensive Case Management)
3. have a terminal medical illness with <3 years expected longevity, or
4. unable to provide informed consent for this study. (Ineligibility to be confirmed based on registry review and Survey Coordinator's assessment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (SF-12) | 3 and 6 months

SECONDARY OUTCOMES:
Bipolar Disorder symptoms (Internal State Scale) | 3 and 6 months
Functioning (WHO-DAS) | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Kilbourne, PhD, Principal Investigator — University of Michigan
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States